CLINICAL TRIAL: NCT03682250
Title: Electrocardiographic Modifications During Spontaneous Hypoglycemic Episodes in Patients with Type 1 Diabetes At High Cardiovascular Risk
Brief Title: Electrocardiographic Modifications and Spontaneous Hypoglycemic Episodes in Type 1 Diabetes
Status: Terminated | Type: Observational
Why Stopped: No one with the qualifications required to analyse the data.
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Other Study IDs: FRYPOT
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with type 1 diabetes with a high cardiovascular risk
  Interventions: Device: FreeStyle Libre Pro; Device: Holter monitor

INTERVENTIONS:
Device: FreeStyle Libre Pro — A FreeStyle Libre Pro will be used to identify hypoglycemic episodes
Device: Holter monitor — A Holter monitor will be used to measure heart's activity

SUMMARY:
The population of type 1 diabetes patients with cardiovascular disease is increasing and this study aims to explore the electrocardiographic changes that are associated with spontaneous hypoglycemia in this type of population. More precisely, this study will investigate if these modifications are of the same nature as those already observed in different populations (patients with type 2 diabetes) to see the pro-arrhythmogenic impact of hypoglycemia in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old;
* Be able to give informed consent;
* Diagnosis of type 1 diabetes for ≥ 6 months;
* Treated with intensive insulin therapy (multiple injections of insulin or insulin pump)

AND EITHER

* A history of CV disease defined as: 1) Established diagnosis of atherosclerotic coronary artery disease (example: previous history of infarction); 2) Previous cerebral Vascular Stroke or Transient Ischemic Accident; 3) Anterior revascularization of the coronary arteries, carotid artery or peripheral arteries; 4) At least one coronary stenosis, carotid artery or lower extremity arteries > 50%; 5) History of symptomatic coronary heart disease confirmed with hospitalization or a positive stress test result or by any cardiac imaging result, or unstable angina with changes observed at the ECG; 6) Asymptomatic cardiac ischemia confirmed by a nuclear imaging test, an exercise test, a dobutamine stress echo; 7) NYHA II-III class chronic heart failure; 8) Amputation of limb or foot due to circulatory insufficiency.
* Or more than 20 years duration of T1D and at least 2 of the following risk factors or associated condition: 1) Chronic renal failure eGFR <60 ml / min / 1.73 m2); 2) Presence of micro or macro-albuminuria (albumin / creatinine ratio > 2); 3) Hypertension or treatment for hypertension; 4) Hyperlipidemia or treatment for hypolipemia; 5) Abdominal obesity (Waist circumference> 94 cm for men and > 80 cm for women); 6) Smoking ; 7) Significant retinopathy (pre-proliferative, proliferating, laser or intravitreous injection); 8) Body mass index > 30 kg /m2; 9) Erectile dysfunction; 10) Left ventricular hypertrophy; 11) Positive family history of early MCAS (H < 55 years old and F < 65 years old)

Exclusion Criteria:

* Definitive criteria: 1) QRS > 120 ms on the baseline ECG; 2) Presence of atrial fibrillation at inclusion; 3) Current intake of any drug that may prolong QT according to the judgment of the investigator and the update of the list available on www.professionsante.com.
* Transient criteria (the patient can be included once the anomaly is corrected): 1) Hypokalemia (< 3.5 mmol/L); 2) Hypocalcemia (ionized calcium < 1.10 mmol/L); 3) Hypomagnesemia (< 0.7 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with type 1 diabetes presenting a high cardiovascular risk
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
QT intervals corrected for heart rate | 48 hours

SECONDARY OUTCOMES:
Percentage of time between 4.0 and 10.0 mmol/L | 48 hours
Percentage of time below 3.5 mmol/L | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No